CLINICAL TRIAL: NCT02258295
Title: Hyaluronate Injection for Lateral Epicondylitis: A Double-blind Randomized Controlled Trial
Brief Title: Hyaluronate Injection for Lateral Epicondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014813CTIL
Record Dates: First submitted 2014-09-14; First posted 2014-10-07 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Tennis Elbow
Keywords: Lateral Humeral Epicondylitis; Tendinitis; Tendinosis; Athletic Injuries; Elbow Joint; Sports Medicine
MeSH Terms: conditions — Tennis Elbow; Tendinopathy; Athletic Injuries | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intragel (Experimental): Intragel (IBSA) has an average size of 800-1200 kDaltons. Intragel will give given with a concentration of 16mg/2cc. Each injection (2cc) injection will be given at baseline, then 2 weeks and 4 weeks from the baseline.
  Interventions: Drug: Intragel
- Saline (Active Comparator): Saline injections will be given similar to the active hyaluronic injections. Each injection (2cc) will be given at baseline, then 2 weeks and 4 weeks from the baseline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Intragel — Intragel has an average molecular weight of 800-1200 kDaltons.
  Other Names: Sinovial; hyaluronate
  Arms: Intragel
Drug: Saline — Saline
  Arms: Saline

SUMMARY:
This proposal is a prospective, randomized, double-blinded study to evaluate the efficacy of hyaluronic acid (HA) injections for chronic lateral epicondylitis (LE). HA has traditionally been used to treat knee osteoarthritis. There are a small number of studies in the literature that suggest that HA injections can be very effective for tendinosis. Although LE has been studied with literally hundreds of articles published, very little treatment has proven to be efficacious. This study will investigate the effectiveness of hyaluronate in treatment of chronic LE. This will include a two arm study with one formulation of HA tested against saline injections as the control.

DETAILED DESCRIPTION:
Patients will be randomized and blinded into one of the two arms. Patients will receive 3 injections total spaced over a 4 week period. After the injections are completed, patients will return for evaluation at 3, 6 and 12 months from the initial injection. A total of 72 patients will be divided into the 2 groups. The questionnaires will be administered by a research assistant blinded to the randomization. Three different outcomes measures will be collected, all patient-oriented including the Patient Rated Tennis Elbow Evaluation (PRTEE), Visual Analog Score (VAS) for pain while at rest and with maximum grip, and the short form Disabilities of the Arm, Shoulder and Hand (quickDASH).

The primary outcome measure will be the VAS for pain at 3 months from the initial injection. All measures will be evaluated at baseline then again at 12 months from the initial injection.

HA formulation will be Intragel (IBSA) which include 2cc with a concentration of 16mg per 2cc. The molecular weight with Intragel averaging 800-1200 kiloDaltons.

The syringes will be coded and the injections blinded. The injections will be given 1cm distal to the lateral epicondyle at the site of maximum tenderness. The needle will be introduced to the depth of the bone then withdrawn 1-2mm. The injection will be given in two locations in and around the point of maximum tenderness.

ELIGIBILITY:
Inclusion Criteria:

* Included will be patients older than 18 years with lateral epicondylitis. The criteria for diagnosis will include pain and tenderness at the lateral epicondyle worse with resisted wrist or finger extension (with the elbow in the extended position).

Exclusion Criteria:

* Excluded will be patients with history of prior elbow surgery, history of fracture or dislocation, known inflammatory or autoimmune disorders, or known hypersensitivity to HA.
* Exclusion will also include a known allergy to birds, feathers or egg products. If the patient has complaints of pain or tenderness on exam in the area of the radial neck, then a component of radial tunnel syndrome will be assumed and these patients will be excluded from study.
* Patients that are pregnant will be excluded.
* Patients with medial epicondylitis
* Prior elbow surgery
* Elbow steroid injection in the past 3 months
* Inflammatory condition, like rheumatoid arthritis or lupus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) for pain with maximum grip. | 3 months from baseline.
  For the (visual analogue score) VAS pain score, patients will be asked to rate their pain after performing a maximum grip using a Jamar hydraulic dynamometer. They will score their pain using the VAS.

SECONDARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation (PRTEE): Change from Baseline to value at 12 | Baseline then 3,6 and 12 months from baseline.
  This is a 15 question validated survey, specific to tennis elbow. It is composed of a pain and function measure. The best score of 0 represents no pain and maximum function.
Visual Analogue Score (VAS) for pain at rest. | Baseline then 3, 6, and 12 months from baseline.
  For this VAS pain score, patients will be asked to rate their pain using the following standard question: "How much pain do you feel when doing an activity that involves gripping such as shaking hands, opening a jar or carrying something?". They will then score their level of pain using the VAS.

OTHER OUTCOMES:
Quick - Disabilities of the Arm, Shoulder and Hand (QuickDASH) | Baseline then 3, 6, and 12 months from baseline.
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.

CONTACTS AND LOCATIONS:
Overall Officials: Gershon Zinger, MD MS, Principal Investigator — Shaare Zedek Medical Center, Jerusalem Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Petrella RJ, Cogliano A, Decaria J, Mohamed N, Lee R. Management of Tennis Elbow with sodium hyaluronate periarticular injections. Sports Med Arthrosc Rehabil Ther Technol. 2010 Feb 2;2:4. doi: 10.1186/1758-2555-2-4. PMID 20205851